CLINICAL TRIAL: NCT05013281
Title: Suprachoroidal Hemorrhage Associated With Pars Plana Vitrectomy
Status: Completed | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TR2021SCH
Record Dates: First submitted 2021-08-11; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Suprachoroidal Hemorrhage (Diagnosis); Pars Plana Vitrectomy
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Suprachoroidal hemorrhage associated with pars plana vitrectomy — SCH has a higher incidence rate after a second intraocular surgery in a vitrectomized eye which is associated with the lack of vitreous support and easier fluctuation of intraocular pressure. SCH associated with PPV is more localized and has a relatively good prognosis; high myopia and aphakic/ pseudophakic eyes are risk factors. Active treatment can effectively improve visual prognosis.

SUMMARY:
To analyze the characteristics, related risk factors, and prognosis of suprachoroidal hemorrhage (SCH) associated with pars plana vitrectomy (PPV).

ELIGIBILITY:
Inclusion Criteria:

* Suprachoroidal hemorrhage associated with pars plana vitrectomy

Exclusion Criteria:

* Patients with eye trauma-related Suprachoroidal hemorrhage were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: any participants who treated with PPV and occured Suprachoroidal hemorrhage with PPV
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
pathogenesis | baseline
  pathogenesis of PPV-related SCH and incidence of PPV-related SCH

SECONDARY OUTCOMES:
vision acuity | up to 7 weeks
  the final vision acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China